CLINICAL TRIAL: NCT04384822
Title: Efficacy of Tai Chi Versus Cognitive Behavioral Therapy for Insomnia (CBT-I) to Treat Chronic Insomnia in Older Adults: A Randomized Controlled Non-inferiority Trial
Brief Title: Efficacy of Tai Chi Versus CBT-I in Treating Chronic Insomnia in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Parco M. Siu, PhD, Associate Professor and Division Head, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 303005RF-002
Record Dates: First submitted 2020-04-03; First posted 2020-05-12 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Chronic Insomnia
Keywords: Clinical Efficacy, Chronic Insomnia, Tai Chi, CBT-I
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcome assessors are unaware of the group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tai Chi Group (Experimental): Subjects will participate in a tai chi program conducted in small groups (10 subjects per group) delivered by qualified instructors, who have experience in teaching tai chi to older adults. The tai chi intervention will be prescribed as a 3-month program with two 1-hour sessions weekly. Tai chi forms will be taught for 2 months followed by 1 month of consolidation. The 24-form simplified Yang-style tai chi will be adopted, as it is the most popular form of tai chi and older adults can manage to learn this simplified form of tai chi within 2-3 months. The instructors will introduce the safety issues, proper training principles, and skills to the subjects in their first class to minimize any avoidable adverse events due to improper skill/practice. The appropriate intensity will be individually determined for each subject by the attending instructors to achieve the training principle of progressive adaptation regarding the exercise intensity.
  Interventions: Behavioral: Tai Chi Group
- CBT-I Group (Active Comparator): Subjects will participate in a conventional CBT-I program conducted in small groups (10 subjects per group) delivered by trained personnel. The CBT-I will be prescribed as a 3-month program with two 1-hour sessions weekly. The CBT-I components will be delivered for 2 months, which is consistent with the duration of the majority of CBT-I treatments, followed by 1 month of consolidation.
  Interventions: Behavioral: CBT-I Group

INTERVENTIONS:
Behavioral: Tai Chi Group — Mind-body exercise intervention
  Arms: Tai Chi Group
Behavioral: CBT-I Group — First-line clinically recommended non-pharmacological treatment of insomnia
  Arms: CBT-I Group

SUMMARY:
Insomnia is common in the older population, over 50% of older adults have sleep complaints, and 20-40% are reported to have insomnia. In HK, 38% of adults have reported insomnia. Insomnia is associated with increased mortality and morbidity. As the worldwide population continues to age, insomnia in older adults will increasingly cause substantial economic burdens on healthcare systems and society.

Cognitive behavioral therapy for insomnia (CBT-I) is currently the first-line clinically recommended non-pharmacological treatment for insomnia in older persons. Our group has been actively studying the health-enhancing effects of tai chi. Tai chi has various health benefits including fall prevention, osteoarthritis management, cardiorespiratory fitness and improvement of sleep. In the present study, the investigators want to validate the clinical effectiveness of tai chi on improving insomnia in older adults. This study aims to exam whether three months of CBT-I or three months of tai chi have similar robust effects in treating insomnia in older adults.

The investigators want to validate the clinical effectiveness of tai chi on improving insomnia in older adults. The CBT-I and tai chi classes will be held twice a week with each lasting for 60 mins. The treatment is three months with 12-month follow-up.

The primary outcome of this study is the insomnia severity index (ISI) score at post-intervention measure, which examining sleep-onset and sleep maintenance difficulties, satisfaction with current sleep pattern, inference with daily functioning.

ELIGIBILITY:
Inclusion Criteria:

1. 50 years or older,
2. ethnic Chinese who can communicate by Cantonese or Mandarin, and
3. fulfill the DSM-5 criteria for chronic insomnia including difficulty in initiating sleep, maintaining sleep or non-restorative sleep, with complaints of impaired daytime functioning, sleep difficulty occurring at least three nights per week present for at least 3 months.

Exclusion Criteria:

1. cannot walk without assistive device (e.g., cane),
2. somatic conditions that limit exercise participation (e.g., limb loss),
3. regular aerobic exercise or mind-body training such as tai chi, yoga, qigong or meditation (>3 times weekly for >60 minutes per session),
4. serious chronic diseases known to affect sleep (e.g., cancer and autoimmune diseases),
5. dementia or use of anti-dementia medication,
6. under treatment for serious diseases known to affect sleep (e.g., cancer chemotherapy),
7. any chronic pain disorders known to affect sleep,
8. untreated sleep disorder including obstructive sleep apnea, periodic leg movement disorder and narcolepsy (screened by questionnaire followed by polysomnographic confirmation in our Co-I's sleep lab, if needed),
9. having current or past CBT-I,
10. shift-worker.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2023-10-27 (Actual); Study Completion 2023-11-02 (Actual)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI) | 3-month follow-up
  ISI will be used to assess the perceived insomnia severity. ISI has seven items examining sleep-onset and sleep maintenance difficulties, satisfaction with the current sleep pattern, interference with daily functioning, noticeable impairment due to sleep problems, degree of distress, and concerns caused by sleep problems. All 160 participants will complete this subjective questionnaire in paper-pencil based manner.
Insomnia Severity Index (ISI) | 15-month follow-up
  ISI will be used to assess the perceived insomnia severity. ISI has seven items examining sleep-onset and sleep maintenance difficulties, satisfaction with the current sleep pattern, interference with daily functioning, noticeable impairment due to sleep problems, degree of distress, and concerns caused by sleep problems. All 160 participants will complete this subjective questionnaire in paper-pencil based manner.

SECONDARY OUTCOMES:
Remission of Chronic Insomnia-Semi-Structured Interview | 3-month follow-up and 15-month follow-up
  The DSM-5 criteria for chronic insomnia will be used to assess the remission of chronic insomnia. All 160 participants will be led by research personnel to complete the brief insomnia questionnaire in a semi-structured interview.
Treatment Response-Insomnia Severity Index (ISI) | 3-month follow-up and 15-month follow-up
  Treatment response is defined as a decrease in the Insomnia Severity Index (ISI) by at least 8 points, which indicates marked improvement or nearly complete or complete remission of insomnia symptoms.
7-day Actigraphy | 3-month follow-up and 15-month follow-up
  A wrist actigraph (wGT3X-BT, Actigraph; a 3-axis accelerometer waterproof watch-like device) that detects movement or lack of movement correlating with wakefulness and sleep, respectively, will be used to objectively estimate sleep. All 160 participants will be instructed to wear an actigraph on the non-dominant wrist for 24 hours per day for 7 days. Actigraphic data will be analyzed by the ActiLifeV6.11.7 software to determine the sleep efficiency.
7-day Sleep Diary | 3-month follow-up and 15-month follow-up
  All 160 participants will be instructed to record their sleep pattern each morning for 7 days using the provided log sheet that records information on bedtime, sleep rising time, total time in bed (TIB), sleep-onset latency (SOL), wake time after sleep onset (WASO), and total sleep time (TST). Sleep efficiency (SE) is estimated as TST/TIB x 100%.
Pittsburgh Sleep Quality Index (PSQI) | 3-month follow-up and 15-month follow-up
  PSQI is a standardized instrument to estimate sleep quantity and quality. There are 19 items that subjectively assess sleep quantity, perceived restfulness, and disturbance of sleep by gathering information on usual bedtime, wake time, time to fall asleep, time of actual sleep, and quality of sleep. All 160 participants will be asked to complete this questionnaire in paper-pencil based manner.
Sleep Medication Record | 3-month follow-up and 15-month follow-up
  The use of sleep aid medications such as narcotics, antihistamines (diphenhydramine), benzodiazepines (e.g., flurazepam, etc), non-benzodiazepine, and benzodiazepine receptor agonists (e.g., zolpidem, etc) with detailed usage information (e.g., drug name, type, dose, and weekly frequency) will be recorded. All 160 participants will be asked to provide the dose and frequency of any sleep medications used by responding to a checklist of all available sleep medications. Data on medication dose and weekly frequency will be presented as the total number of lowest recommended dose (LRD) in 7 days.
Quality of Life by Standard SF-12 Health Survey (SF12v2) | 3-month follow-up and 15-month follow-up
  The Chinese version SF-12, derived from the SF-36, will be used to measure health-related quality of life. There are 12 items assessing physical functioning, emotional and mental health, bodily pain, general health, vitality, and social functioning, with higher overall scores indicating a better quality of life. The Chinese version SF- 12 has been validated in the Hong Kong Chinese population. All 160 participants will be asked to complete this questionnaire in paper-pencil based manner.
Mental Health by Hospital Anxiety and Depression Scale (HADS) | 3-month follow-up and 15-month follow-up
  Hospital Anxiety and Depression Scale (HADS) will be used to evaluate the severity of depression and anxiety. This 7-item questionnaire has an overall score ranging from 0 to 21 (with subscales for both anxiety and depression), with a higher score indicating more severe symptoms. All 160 participants will be asked to complete this questionnaire in paper-pencil based manner.
Balance and Lower Extremity Function by Short Physical Performance Battery (SPPB) | 3-month follow-up and 15-month follow-up
  SPPB will be used to assess balance and lower extremity function. SPPB includes repeated timed chair stands, timed standing balance (with feet in parallel, semi-tandem, and tandem positions), and a 4-meter walk to measure the usual gait speed. These outcomes will objectively validate the receipt of the tai chi intervention based on the known benefits of tai chi on balance and lower extremity performance. The investigators will assess the balance and lower extremity function during the baseline measurement.
Adverse Events | 3-month follow-up and 15-month follow-up
  Adverse events (such as injuries related to interventions or not) will be closely monitored and recorded through regular surveys by instructors and research personnel, and by voluntary reports from the subjects. Subjects with sustained serious adverse events that affect their daily function will terminate the study, but their data will be included in our ITT analyses.
Habitual Physical Activity | 3-month follow-up and 15-month follow-up
  Potential confounding factors including changes in habitual physical activity will be monitored. The habitual physical activity will be assessed by the international physical activity questionnaire and 7-day actigraph.
Dietary Intake | 3-month follow-up and 15-month follow-up
  The diet will be assessed by a 3-day food diary. The research personnel will explain how to fill a 3-day food diary and all 160 participants will be asked to complete these 3 measurements

CONTACTS AND LOCATIONS:
Overall Officials: Ming Fai P. Siu, PhD, Principal Investigator — School of Public Health, The University of Hong Kong
Locations (1):
- School of Public Health, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The data of individual participants that underlie the results reported in this trial, after de-identification including text, tables, figures, and appendices, as well as study protocol and statistical analysis plan, will be shared after 3 months of study publication. Data will be shared with researchers who provide a methodologically sound proposal for academic purposes. Proposals should be directed to pmsiu@hku.hk to gain access and for data request, a data-access agreement needs to be signed.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months and ending 3 years following the publication of the article
Access Criteria: Data will be shared with researchers who provide a methodologically sound proposal for academic purposes. Proposals should be directed to pmsiu@hku.hk to gain access and for data request, a data-access agreement needs to be signed.

REFERENCES:
- [Derived] Siu PM, Yu DJ, Yu AP, Recchia F, Li SX, Chan RN, Fong DY, Chan DK, Hui SS, Chung KF, Woo J, Wang C, Irwin MR. Tai chi or cognitive behavioural therapy for treating insomnia in middle aged and older adults: randomised non-inferiority trial. BMJ. 2025 Nov 26;391:e084320. doi: 10.1136/bmj-2025-084320. PMID 41297969